CLINICAL TRIAL: NCT00026416
Title: Phase II Study of Low-Dose Interferon Alfa 2B (Schering Plough) Plus Thalidomide (Celgene) for Patients With Resected High-Risk Soft Tissue Sarcoma
Brief Title: Interferon Alfa and Thalidomide in Treating Patients With Soft Tissue Sarcoma or Bone Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069028; CPMC-IRB-13887; NCI-G01-2024
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-10

CONDITIONS: Sarcoma
Keywords: stage III adult soft tissue sarcoma; localized osteosarcoma; metastatic osteosarcoma; stage II adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Interferon-alpha; Thalidomide; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: thalidomide
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Interferon alfa may interfere with the growth of cancer cells. Combining interferon alfa and thalidomide may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining interferon alfa and thalidomide in treating patients who have undergone surgery for soft tissue sarcoma or bone sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of interferon alfa and thalidomide, in terms of time to disease progression, in patients with surgically resected high-risk soft tissue sarcoma or bone sarcoma.
* Determine the incidence of metastatic disease and overall survival in patients treated with this regimen.
* Determine the clinical and laboratory toxic effects and the tolerability of this regimen in these patients.

OUTLINE: Patients receive interferon alfa subcutaneously three times a week on weeks 1-60 and oral thalidomide once daily on weeks 13-60 in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 weeks for at least 2 years.

PROJECTED ACCRUAL: A total of 20-48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary or metastatic soft tissue sarcoma or bone sarcoma at high risk of recurrence

  * Grade III-IV tumor greater than 8 cm
  * Grade III-IV primary tumor greater than 5 cm with positive surgical margins
  * Grade III-IV primary tumor greater than 5 cm with distant metastases resected within 1 year of primary surgery
* No more than 8 weeks since prior surgical resection of primary or metastatic disease
* Ineligible for other high priority national or institutional study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count greater than 70,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT or SGPT less than 3 times upper limit of normal (ULN)*
* Alkaline phosphatase less than 3 times ULN*
* No decompensated liver disease
* No autoimmune hepatitis
* No coagulation disorders NOTE: * Unless due to metastatic disease

Renal:

* Creatinine normal

Cardiovascular:

* No history of severely debilitating cardiovascular disease
* No unstable angina
* No uncontrolled congestive heart failure
* No thrombophlebitis

Pulmonary:

* No history of severely debilitating pulmonary disease
* No chronic obstructive pulmonary disease
* No pulmonary embolism

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception for 4 weeks before, during, and for 4 weeks after study
* No acute infection requiring systemic antibiotics
* No prior hypersensitivity to interferon alfa or any component of the injection
* No diabetes mellitus prone to ketoacidosis
* No severe myelosuppression
* No history of autoimmune disease
* No pre-existing thyroid abnormalities with thyroid function that cannot be maintained in the normal range
* No clinically significant retinal abnormalities
* No other serious medical or psychiatric illness that would preclude study
* No prior malignancy except curatively treated carcinoma in situ of the cervix or skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior systemic chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Taub, MD, PhD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States